CLINICAL TRIAL: NCT05703048
Title: The Effect of Esmolol Versus Dexmedetomidine on Postoperative Pain Control in Endoscopic Sinus Surgery: A Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Faheem, Assistant professor of anesthesiology, intensive care, and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: esmolol versus dexmedetomidine
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Patient's Satisfaction; Depth of Anesthesia
Keywords: postoperative pain; emergence of aneasthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — esmolol esterase; esmolol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: In group A (dexmedetomidine group): 35 patients will be received dexmedetomidine (Precedex; Abbott Laboratories, North Chicago, Illinois, USA) (vial = 2 ml) 100 mcg/ml at bolus dose of 1 mcg /kg slowly infused over 10 min, then continuous infusion by a rate of 0. 5 mcg /kg/h., infused by a syringe pump. infusion stopped immediately upon extubation.
  In group B (Esmolol group): 35 patients will be received i.v. received a loading dose of esmolol 0.5 mg/kg in 30 mL isotonic saline in the IV line, followed by an IV infusion of esmolol 0.05 mg/kg/min. infusion stopped immediately upon extubation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer system will be used for randomization by creating a list of number each number referred to one of the two groups. Block randomization will be used to ensure equality of the groups. Each number will be sealed in an opaque envelope. Then, each patient will be asked to choose one of the envelopes and give it to an anesthesiologist who compared it to the computer-generated list and hence assigned her to one of the two groups. The anesthesiologist, participant and outcomes Assessor will be blinded to the collected data until the end of the study and administered the medication.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Experimental): 35 patients will be received dexmedetomidine (Precedex; Abbott Laboratories, North Chicago, Illinois, USA) (vial = 2 ml) 100 mcg/ml at bolus dose of 1 mcg /kg slowly infused over 10 min, then continuous infusion by a rate of 0. 5 mcg /kg/h., infused by a syringe pump. infusion stopped immediately upon extubation.
  Interventions: Drug: Dexmedetomidine
- Esmolol group (Active Comparator): 35 patients will be received i.v. received a loading dose of esmolol 0.5 mg/kg in 30 mL isotonic saline in the IV line, followed by an IV infusion of esmolol 0.05 mg/kg/min. infusion stopped immediately upon extubation.
  Interventions: Drug: Esmolol Esterase

INTERVENTIONS:
Drug: Esmolol Esterase — 35 patients will be received i.v. received a loading dose of esmolol 0.5 mg/kg in 30 mL isotonic saline in the IV line, followed by an IV infusion of esmolol 0.05 mg/kg/min. infusion stopped immediately upon extubation.
  Other Names: Esmolol
  Arms: Esmolol group
Drug: Dexmedetomidine — 35 patients will be received dexmedetomidine (Precedex; Abbott Laboratories, North Chicago, Illinois, USA) (vial = 2 ml) 100 mcg/ml at bolus dose of 1 mcg /kg slowly infused over 10 min, then continuous infusion by a rate of 0. 5 mcg /kg/h., infused by a syringe pump. infusion stopped immediately upon extubation.
  Arms: dexmedetomidine group

SUMMARY:
Hypotensive techniques are associated with certain disadvantages. Hence, anesthesiologists are still in search of drugs with fewer side effects.

Various drugs such as high-concentration volatile anesthetics, magnesium sulfate, remifentanil, clonidine, calcium channel blockers, tranexamic acid, intravenous nitroglycerin, and sodium nitroprusside have been evaluated to control blood pressure and decrease blood loss during surgery, thereby improving the surgical field quality.

Opioids are the mainstay of treatment for perioperative pain, but their administration increases the incidence of respiratory complications, slows down normal gastrointestinal motility, and prolongs hospital stay. With the development of enhanced recovery after surgery (ERAS), reducing the use of opioids in the perioperative period has become the common goal of anesthesiologists. The dosage of opioids should be strictly controlled whenever possible, which should not only meet the needs of analgesia perioperatively, but also minimize the incidence of adverse reactions.

Opioid-free anesthesia (OFA) represents a step forward in anesthetic practice as it potentially spares the use of opioids by administrating nonopioid agents and adjuncts. The rationale to propose OFA is based on the aim to avoid the negative impact of intraoperative opioids on a patient's postoperative outcomes.

Several studies showed that β adrenergic receptor antagonists withhold the upsurge of catecholamines circulating in blood which induced by surgery, as well as having analgesic sparing effect itself. Esmolol is an ultrashort acting β1 blocking drug that has been uncovered to own opioid-sparing effects likely due to resemblances in its structure with local anesthetic agents. Esmolol's short course of action and titrability offer it as an attractive drug to use, although the mechanism of action of its analgesic effect has yet to be established.

Dexmedetomidine hydrochloride is a specific alpha-2 adrenoreceptor agonist that has intrinsic analgesic and sedative properties coupled with anxiolytic and sympatholytic effects. It minimizes the hemodynamic and neuroendocrine responses to anesthesia and surgery by suppressing the sympathetic tone. This hemodynamic stability can improve the surgical outcome as well as both patient and surgeon satisfaction. Dexmedetomidine accompanied by other anesthetics causes a controlled reduction in blood pressure and heart rate and improves the quality of the surgical field.

Alpha-2 adrenergic agonists (dexmedetomidine) have pharmacologic characteristics (sedation, hypnosis, anxiolysis, sympatholytic, and analgesia) that make them suitable as adjuvants to multimodal analgesia.

Their anti-nociceptive effect is attributed to the stimulation of a2- adrenoceptors located in the central nervous system. Dexmedetomidine is a highly selective and potent a2-adrenoceptor agonist. Its intrathecal administration leads to anti-nociceptive effects, although it does have some undesired side effects (e.g., hypotension, bradycardia, and sedation).

DETAILED DESCRIPTION:
This randomized prospective study will be carried out in Tanta university hospital in the ENT surgery department on 70 Patients with American Society of Anesthesiologists (ASA) Physical Status Class I &II, aged > 18 years and scheduled for FESS.

After approval from the institutional ethics committee, informed consent will be obtained from all participants parents in this research.

A computer system will be used for randomization by creating a list of number each number referred to one of the two groups. Block randomization will be used to ensure equality of the groups. Each number will be sealed in an opaque envelope. Then, each patient will be asked to choose one of the envelopes and give it to an anesthesiologist who compared it to the computer-generated list and hence assigned her to one of the two groups. The anesthesiologist, participant and outcomes Assessor will be blinded to the collected data until the end of the study and administered the medication.

The patients will be taken to the preoperative room 30 minutes before the operation. Patients are randomly divided into two groups ( 35 each):

In group A (dexmedetomidine group): 35 patients will be received dexmedetomidine (Precedex; Abbott Laboratories, North Chicago, Illinois, USA) (vial = 2 ml) 100 mcg/ml at bolus dose of 1 mcg /kg slowly infused over 10 min, then continuous infusion by a rate of 0. 5 mcg /kg/h., infused by a syringe pump. infusion stopped immediately upon extubation.

In group B (Esmolol group): 35 patients will be received i.v. received a loading dose of esmolol 0.5 mg/kg in 30 mL isotonic saline in the IV line, followed by an IV infusion of esmolol 0.05 mg/kg/min. infusion stopped immediately upon extubation.

In all groups, Anesthesia induction with propofol 1% 2 mg/kg, lidocaine 1mg/kg and rocuronium 0.5 mg/kg. No supplemental opioids will be used during the surgery.

The airway will be secured with an appropriate size tracheal tube. Anesthesia will be maintained using a mixture of O2 and air in a ratio of 1:1 mixture with 2% sevoflurane (MAC adjusted to keep the BIS index between 40 and 60). The ventilator settings will be adjusted to maintain normocapnia. Intraoperative monitoring included electrocardiogram, pulse oximetry, blood pressure, end tidal carbon dioxide, end tidal sevoflurane concentration (Et.Sev), and temperature. Fluids will be given at 10 ml/kg/h in the form of dextrose 5% and normal saline at a ratio of 1:1.

Controlled hypotension will be defined as mean arterial pressure (MAP) of 55-65 mmHg. Any intraoperative or postoperative complications, such as excessive hypotension (MAP <50 mmHg), hypertension (MAP >10% of baseline), need of additional hypotensive agents or vasopressors, tachycardia, bradycardia, bronchospasm, arrhythmias or delayed recovery will be noted. Rescue antihypertensive agent will be nitroglycerine and the patients requiring it will be excluded from the study. In the case of a higher MAP leading to excessive bleeding in the surgical field, a nitroglycerin infusion will be started at a dose of 0.5 μg/kg/min. If the arterial blood pressure fell to less than 30% of the baseline MAP, first an intravenous fluid infusion will be used to correct the blood pressure, with a bolus ephedrine dose of 5 mg being administered if the former will be insufficient.

Bradycardia will be generally self-limiting and will be corrected spontaneously after stopping infusion of esmolol if required. If the heart rate dropped to less than 44 beats per minute, atropine 0.6 mg will be given as a bolus. All prescribed drugs will be recorded.

The end of the operation will be defined as when the surgeon and the assistant surgeon performed the dressing and announced the completion of surgery. At this time, all anesthetics will be discontinued, and the patient will be ventilated with 100% oxygen. After the return of respiratory signs or any movements, the patients will be given neostigmine (0.05 mg/kg IV) and atropine (0.02 mg/kg IV). Once the patient's tidal volume reached two-thirds of the expected value and the patient would obey orders, he or she will be extubated. The bed of each patient will be situated in the head-up (10 degrees) position. When an Aldrete score of ≥ 9 will be achieved, patients will be discharged from the PACU.

Postoperative pain management included oral acetaminophen 500 mg\6 h as a fixed dose.

Blindness For injection of medication ahead of anesthesia induction, identical syringes (in equal volumes) containing three used drugs and normal saline will be prepared by a physician not involved in the research based on a table provided by the statistician. The syringes will be delivered to the treating physician, who injected them at the specified time without knowing the type of drug. All patients and physicians will be unaware of the type of drug and study group.

Measurements:

1. A demographic information, including age, sex and weight of the patient, and duration of the operation will be recorded.
2. Monitoring of the depth of anesthesia will be conducted by the Bispectral Index (BIS). The BIS will be measured by a BIS monitor (BIS; Aspect Medical Systems, Newton, Massachusetts) which then calculates the depth of anesthesia by the BIS as a number. A BIS less than 40 demonstrates very deep anesthesia, 40-60 means surgical anesthesia, 61-80 means light anesthesia, more than 81 demonstrates sedation, and 100 shows full awareness.
3. Assessing VAS score for pain will be done by the blinded investigator in the PACU (on arrival, 1 h) and in surgical ward (at 6 h, 12 h and 24 h). IV 5 mg morphine will be given if VAS score exceeded 4.
4. The patients' behaviour during emergence from anesthesia and in the PACU will be rated the 6-point RSS scores (1 = patient anxious and restless, 2 = cooperative and awake, 3 = responding to verbal commands, 4 = responding to mild stimulus, 5 = responding to deep stimulus, 6 = no.
5. Percentage of patients receiving rescue opioids.
6. Patient's satisfaction will be also evaluated depending on a 5-point Likert scale as follow: (1-very unsatisfied, 2-unsatisfied, 3-unsure, 4-satisfied, and 5-very satisfied).
7. These included increased sleepiness (Ramsay sedation scale (RSS) score > 3), respiratory depression (SpO2 < 90% in room air or respiratory rate < 8/min).
8. Subjective assessment of the surgical field for bleeding will be carried out by the surgeon according to category scale adapted from Fromme et al., Category scale values of 2 and 3 for the surgical field will be considered as ideal. The blood will be sucked in a preheparinized suction canister. The amount of blood loss will be calculated from the fluid volume of the suction canister (V), the Hb concentration of the suction canister, and the patient's mean Hb concentration at the beginning and end of surgery (Hbm) using the following equation:
9. Blood loss (mL) = Hb (gdL/1) × V (mL)/Hbm (g/dL).
10. The recovery time (time between the cessation of maintenance anesthetics and eye-opening) by the minute.
11. Time to extubation (time from the discontinuation of sevoflurane to the removal of endotracheal tube) by minute.
12. Length of staying in PACU will be defined as the time between arrival and discharge time will be measured. using Aldrete scale, a score of 9 or greater allows the patient to leave the postanesthesia unit.
13. Frequency of nausea, vomiting, on a four point scale (1 = no nausea, 2 = mild nausea, 3 = severe nausea, 4 = retching and/or vomiting),and pruritis during the first 24 hours postoperatively. Subjects experiencing nausea or vomiting received ondansetron 0.15 mg/kg iv every six hours as needed. PONV grade 3 & 4 will be treated with metoclopramide 10 mg IV.
14. The mean arterial pressure (MAP) and heart rate (HR) will be recorded at entering the room (T1), after loading dosage (T2), after anesthesia induction (T3), 1 min after intubation (T4), 5 min after skin cutting (T5), 1h after skin cutting (T6), 2h after skin cutting (T7) and 5min after extubation (T8), respectively.
15. Level of sedation: The level of sedation will be evaluated with the Richmond Agitation Sedation Scale (RASS). This scale ranges from a score of -5 (unarousable) to +4 (intense agitation) in PICU.
16. The incidences of intubation and extubation response will be recorded separately. Intubation response will be considered to have occurred when MAP or HR at 5 minutes after intubation exceeds 15% or more than that at 5 minutes after induction of anesthesia (before intubation). At the same time, when the MAP or HR at 5 minutes after extubation will be 15% or higher than that at 5 minutes before spontaneous breathing occurred before extubation, it will be considered as extubation response.
17. Surgeon satisfaction with surgical field quality: This will be evaluated according to the surgeon's opinion using the Likert scale below:

    * Score 1 (very poor): Uncontrollable bleeding.
    * Score 2 (poor): Severe bleeding requiring repeated suctioning, with the quality of the field collapsing immediately after suctioning.
    * Score 3 (satisfactory): Moderate bleeding requiring intermittent suctioning.
    * Score 4 (good): Partial bleeding, sometimes requiring suctioning; the quality of the surgical field will be good.
    * Score 5 (excellent): No bleeding/bloodless field; the surgery field will be excellent.

ELIGIBILITY:
Inclusion Criteria:

* 70 patients with American Society of Anesthesiologists (ASA) Physical Status Class I&II, aged > 18 years. and scheduled for FESS.

Exclusion Criteria:

* 1. The patients on β-blockers and cardiovascular active drugs 2. History of neuromuscular disorder, diabetic neuropathy, pregnancy 3. Prolonged QT interval and ventricular arrhythmia, specifically a pre-disposition to bradycardia or conduction abnormalities, cyanotic cardiac disease, and use of medications that would increase the risk of bradycardia.

  4. Current (Within the last 30 days) opioid use for pain control as sickle cell disease, substance abuse or benzodiazepine addiction 5. History of end stage hepatic, renal, diabetes mellitus, and bleeding disorders, 6. Allergy and hypersensitivity to the drugs used in the study 7. Excessive use of analgesics/non-steroidal anti-inflammatory drugs 8. Morbid obesity (body mass index (BMI) > 40) 9. A positive history of motion sickness, women who had a history of nausea and vomiting before menstruation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
opioid (morphine) consumption up to 24 hours after end of the surgery. | first 24 hs following surgery.
  opioid (morphine) consumption up to 24 hours after end of the surgery.

SECONDARY OUTCOMES:
visual analog scale (VAS) score for pain ( maximum score was 10 which mean sever pain and least score was 0 which mean no pain) | in the PACU at admission
  VAS score for pain will be done by the blinded investigator in the PACU at admission
visual analog scale (VAS) score for pain ( maximum score was 10 which mean sever pain and least score was 0 which mean no pain) | in the PACU at one hour postoperative
  VAS score for pain will be done by the blinded investigator in the PACU at one hour postoperative
visual analog scale (VAS) score for pain ( maximum score was 10 which mean sever pain and least score was 0 which mean no pain) | in the PACU at 6 hours in surgical ward
  VAS score for pain will be done by the blinded investigator at 6 hours in surgical ward
visual analog scale (VAS) score for pain ( maximum score was 10 which mean sever pain and least score was 0 which mean no pain) | in the PACU at 12 hours in surgical ward
  VAS score for pain will be done by the blinded investigator at 12 hours in surgical ward
visual analog scale (VAS) score for pain ( maximum score was 10 which mean sever pain and least score was 0 which mean no pain) | in the PACU at 24 hours in surgical ward
  VAS score for pain will be done by the blinded investigator at 24 hours in surgical ward

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tantan University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No